CLINICAL TRIAL: NCT01098253
Title: Integrating Depression Services Into Type 2 Diabetes Mellitus Management
Brief Title: Integrating Depression Services Into DM Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Hillary Bogner, MD MSCE/ Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-09-CR-07
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus; Depression
Keywords: adherence; diabetes mellitus; depression; primary health care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adherence Intervention (Experimental): Factors affecting adherence to oral hypoglycemic agents and antidepressants were addressed using a problem solving process.
  Interventions: Behavioral: Adherence Intervention
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Adherence Intervention — Factors affecting adherence are addressed using a problem solving process.
  Arms: Adherence Intervention

SUMMARY:
The goal of this proposal is to integrate depression services into improving adherence for oral hypoglycemic agents so that a single program can assist patients. The investigators hypothesized that patients in the intervention would demonstrate improved adherence to patients' oral hypoglycemic agents and antidepressants as well as improved clinical outcomes.

DETAILED DESCRIPTION:
Many older patients do not take their medications for Type 2 diabetes mellitus (DM) as prescribed by their physician. Depression is common among patients with Type 2 DM and may be the reason why patients do not take their medications as prescribed. A program in which Type 2 DM and depression are treated together in primary care would improve the health of older patients with both Type 2 diabetes and depression and would be practical in real world practices with competing demands for limited resources. There is an urgent need for research that can bring potentially life-extending strategies to older patients with both diabetes and depression. People can better control their Type 2 DM if they treat their depression and the same strategies can be used to help patients take their medications for both conditions. In this program patients were involved in identifying problems with taking their medicines and working on solutions. The aims of this program were to improve how patients take their medications for Type 2 DM and depression as well as blood glucose control and symptoms of depression over 3 months. To see whether this program works the investigators compared the results of patients receiving this program to those who do not receive the program. Findings may lead to the development of other programs in which depression and chronic medical conditions are treated together.

ELIGIBILITY:
Inclusion Criteria:

* 30 years and older
* a current diagnosis of Type 2 DM
* current prescription for an oral hypoglycemic agent
* current prescription for an antidepressant
* able to communicate in English
* willing to give informed consent.

Exclusion Criteria:

* inability to give informed consent
* significant cognitive impairment at baseline (Mini-Mental State Examination (MMSE) <21)
* residence in a care facility that provides medications
* unwillingness or inability to use the Medication Event Monitoring System

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillary R. Bogner, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from three primary care practices in Philadelphia, Pennsylvania. The protocol was approved by the University of Pennsylvania Institutional Review Board. From April 2010 to April 2011, patients were identified and enrolled.
Pre-assignment Details: This trial consisted of two phases: the run-in phase and the randomized controlled trial phase. The purpose of the 2-week run-in phase was to collect pre-intervention adherence rates for all patients.
Groups:
- Integrated Care Intervention: We carried out an integrated care intervention in which the integrated care manager collaborated with physicians to offer education to patients, guideline-based treatment recommendations, and to monitor adherence and clinical status.
Period: Overall Study
Arm/Group | Integrated Care Intervention | Usual Care
Started | 94 | 88
Completed | 92 | 88
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Care Intervention | Usual Care | Total
Number analyzed (Participants) | 94 | 88 | 182
Age Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (9.4) | 57.1 (9.6) | 57.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 58 | 122
  Male | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  United States | 94 | 88 | 182

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C
Description: HbA1c levels will be obtained in accordance with ADA guidelines (1) employing the in2it A1C Analyzer. The Analyzer offers accurate point of care HbA1c testing. Point of care testing using this device has acceptable precision and agreement in comparison with laboratory services
Time Frame: 3 months
Population: Analysis proceeded at the patient level and patients were analyzed according to the treatment to which they were randomized (intent-to-treat).
Measure: Number; unit: Percentage of participants with HbA1c <7
Arm/Group | Integrated Care Intervention | Usual Care
Number analyzed (Participants) | 92 | 88
Percentage of participants with HbA1c <7 | 60.9 (1.8) | 35.7 (1.9)

2. Secondary Outcome: Nine Item Patient Health Questionnaire (PHQ-9)
Description: Depressive symptoms were measured using the nine-item Patient Health Questionnaire (PHQ-9). PHQ-9 scored on a range from 0 to 27, where lower scores represent fewer depressive symptoms.
Time Frame: 3 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants with PHQ-9 <5
Arm/Group | Integrated Care Intervention | Usual Care
Number analyzed (Participants) | 92 | 88
Percentage of participants with PHQ-9 <5 | 58.7 | 30.7

ADVERSE EVENTS:
Arm/Group | Integrated Care Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/88
Other Adverse Events (participants affected / at risk) | 0/94 | 0/88

LIMITATIONS AND CAVEATS:
Our primary care sites might not be representative of most primary care practices. Patients in the usual care group did not have the same number of in person contacts as those in the integrated care intervention to control for attention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No